CLINICAL TRIAL: NCT00699725
Title: Compliance of Gastroprotection Treatment in the Prevention of Gastrointestinal Risk in Non-Steroidal Anti-inflammatory Drug (NSAID) Using Patients
Brief Title: Adherence to Gastro-protection in Non-steroidal Anti-inflammatory Drug (NSAID) Using Patients
Acronym: GADES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Mercedes Muñoz, PhD, Local MC GI Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GES-DUM-2008/2
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Compliance; Gastroprotector Therapy; Risk Factors
Keywords: Compliance; gastroprotector therapy; NSAID; risk factors
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: NSAID patients with risk factors treated with gastroprotective drugs

SUMMARY:
Prospective multicentric study to evaluate the compliance of gastroprotective treatment in NSAID patients at risk of GI complications. Secondary objectives: To identify the factors associated to treatment compliance (both NSAID and PPI), to evaluate the relationship between compliance and NSAID-associated GI events

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients consulting to the specialized care clinics who have been prescribed NSAID and gastroprotection for at least 15 days following standard clinical practice.

Exclusion Criteria:

* Any gastroprotective treatment prescribed for other condition than NSAID-related gastrointestinal event prevention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending secondary care clinics who are prescribed NSAID and gastroprotection for at least 15 days following standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adherence to gastroprotection treatment | End of follow-up (3-5 weeks)

SECONDARY OUTCOMES:
Identify factors associated with treatment compliance | End of follow-up
Evaluate the relationship among GI events and treatment compliance | End of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Javier Zapardiel, Study Chair — AstraZeneca Spain Medical Dept
Locations (128):
- Spain (128):
  - Research Site, Vitoria-Gasteiz, Alava
  - Research Site, Albacete, Albacete
  - Research Site, Alacant / Alicante, Alicante
  - Research Site, Alcoy, Alicante
  - Research Site, Elda, Alicante
  - Research Site, Elx / Elche, Alicante
  - Research Site, La/villajoyosa Vila Joiosa, Alicante
  - Research Site, Orihuela, Alicante
  - Research Site, San Bartolomé, Alicante
  - Research Site, San Vicent del Raspeig, Alicante
  - Research Site, Almería, Almeria
  - Research Site, El Ejido, Almeria
  - Research Site, Huercal Overa, Almeria
  - Research Site, Ávila, Avila
  - Research Site, Badajoz, Badajoz
  - Research Site, Don Benito, Badajoz
  - Research Site, Zafra, Badajoz
  - Research Site, Manacor, Balearic Islands
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Barcelona
  - Research Site, Barcelona, Barcelona
  - Research Site, Castelldefels, Barcelona
  - Research Site, Cornellà de Llobregat, Barcelona
  - Research Site, El Hospitalet de Llobregat, Barcelona
  - Research Site, Granollers, Barcelona
  - Research Site, Manresa, Barcelona
  - Research Site, Martorell, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Sant Boi de Llobregat, Barcelona
  - Research Site, Torrebonica, Barcelona
  - Research Site, Viladecans, Barcelona
  - Research Site, Burgos, Burgos
  - Research Site, Cáceres, Caceres
  - Research Site, Coria, Caceres
  - Research Site, Navalmoral de la Mata, Caceres
  - Research Site, Plasencia, Caceres
  - Research Site, Algeciras, Cadiz
  - Research Site, Cadiz, Cadiz
  - Research Site, El Puerto de Santa María, Cadiz
  - Research Site, Jerez de la Frontera, Cadiz
  - Research Site, Torrelavega, Cantabria
  - Research Site, Castellon, Castellon
  - Research Site, Vinaròs, Castellon
  - Research Site, Puertollano, Ciudad Real
  - Research Site, Valdepe�as, Ciudad Real
  - Research Site, Cabra, Cordoba
  - Research Site, Córdoba, Cordoba
  - Research Site, Puente-Genil, Cordoba
  - Research Site, Cuenca, Cuenca
  - Research Site, Almu�ecar, Granada
  - Research Site, Granada, Granada
  - Research Site, Guadix, Granada
  - Research Site, Motril, Granada
  - Research Site, Guadalajara, Guadalajara
  - Research Site, Mendaro, Guipuzcoa
  - Research Site, Tolosa, Guipuzcoa
  - Research Site, Huelva, Huelva
  - Research Site, Jaén, Jaen
  - Research Site, Linares, Jaen
  - Research Site, Úbeda, Jaen
  - Research Site, A Coru�a, La Coru�a
  - Research Site, Ferrol, La Coru�a
  - Research Site, Oleiros (ribeira), La Coru�a
  - Research Site, Santiago de Compostela, La Coru�a
  - Research Site, Calahorra, La Rioja
  - Research Site, Logro�o, La Rioja
  - Research Site, Las Palmas de Gran Canaria, Las Palmas
  - Research Site, Puerto del Rosario, Las Palmas
  - Research Site, Telde, Las Palmas
  - Research Site, León, Leon
  - Research Site, Lleida, Lerida
  - Research Site, Burela de Cabo, Lugo
  - Research Site, Foz (casco Urbano), Lugo
  - Research Site, Lugo, Lugo
  - Research Site, Monforte (casco Urbano), Lugo
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Aranjuez, Madrid
  - Research Site, El Escorial, Madrid
  - Research Site, Getafe, Madrid
  - Research Site, Leganés, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, Móstoles, Madrid
  - Research Site, Fuengirola, Malaga
  - Research Site, Marbella, Malaga
  - Research Site, Málaga, Malaga
  - Research Site, Melilla, Melilla
  - Research Site, Cartagena, Murcia
  - Research Site, Cieza, Murcia
  - Research Site, El Palmar (el Palmar), Murcia
  - Research Site, Murcia, Murcia
  - Research Site, Santiago de la Ribera, Murcia
  - Research Site, Elcano, Navarre
  - Research Site, Estella-Lizarra, Navarre
  - Research Site, Pamplona, Navarre
  - Research Site, Tudela, Navarre
  - Research Site, Ourense, Orense
  - Research Site, Verín, Orense
  - Research Site, Pontevedra, Pontevedra
  - Research Site, Vigo, Pontevedra
  - Research Site, Vilagarcía de Arousa, Pontevedra
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Murias (mieres), Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Ria�o (langreo), Principality of Asturias
  - Research Site, Castilleja de la Cuesta, Sevilla
  - Research Site, Seville, Sevilla
  - Research Site, Tarragona, Tarragona
  - Research Site, Arona, Tenerife
  - Research Site, Bre�a Alta, Tenerife
  - Research Site, La Orotava, Tenerife
  - Research Site, San Cristóbal de La Laguna, Tenerife
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, Talavera de la Reina, Toledo
  - Research Site, Toledo, Toledo
  - Research Site, Algemesí, Valencia
  - Research Site, Alzira, Valencia
  - Research Site, Port de Sagunt, Valencia
  - Research Site, Requena, Valencia
  - Research Site, Sueca, Valencia
  - Research Site, Torrent, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Xàtiva, Valencia
  - Research Site, Bilbao, Vizcaya
  - Research Site, Galdakao, Vizcaya
  - Research Site, Zamora, Zamora
  - Research Site, Calatayud, Zaragoza
  - Research Site, Zaragoza, Zaragoza